CLINICAL TRIAL: NCT03374839
Title: Combined Therapy of Nivolumab and Adoptive T Cell Therapy in Metastatic Melanoma Patients: Pilot Study Phase I/II
Brief Title: Combined Therapy of Nivolumab and Adoptive T Cell Therapy in Metastatic Melanoma Patients
Acronym: Nivo-TIL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0247
Record Dates: First submitted 2017-11-29; First posted 2017-12-15 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Toll-Like Receptor 1; Interleukin-2; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIL + IL-2 + Nivolumab (Experimental): A first cohort of 3 patients will be done to ensure that the combined treatment (TIL + IL-2 + Nivolumab) would not cause severe autoimmunity pathologies.
  For this first cohort, a dose of 0.5 billion of TILs per injection will be administered. After the opinion of the Data and Safety Monitoring Committee (DSMC), the sponsor will make the decision of the second cohort of 8 patients who will receive between 1 and 20 billion of TIL.
  Interventions: Drug: TIL + IL-2 + Nivolumab

INTERVENTIONS:
Drug: TIL + IL-2 + Nivolumab — The patients will receive Nivolumab (at a dose of 3 mg per kilogram of body weight) every 2 weeks from day0 until week52.
  Two TIL (Tumor Infiltrating Lymphocytes) injections will be performed: at week 14 and at week 18.
  The TIL injections are systematically followed by subcutaneous injections of Proleukin® (IL-2) at a concentration of 6 million international unit (IU) per day for 5 days.

SUMMARY:
To improve the efficacy of immunotherapy for cancer, recent studies focused on specific targets to redirect the immune network toward eradicating a variety of tumors and ameliorating the self-destructive process.

A clinically relevant immune escape mechanism in melanoma is the activation of the Programmed cell Death-1 (PD-1) receptor on infiltrating T cells. By blocking PD-1 receptors with anti-PD-1 monoclonal antibodies (mAbs), T-cells are unaffected by the PD-L1 expressed on tumor cells and the patients T cells are free to respond to melanoma antigens and attack tumor cells. So the objective of this trial is to evaluate the safety and the efficacy of a combined therapy Nivolumab and adoptive T cell therapy in metastatic melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old with a weight ≥ 40 kg
* Patients must have signed informed consent
* Patients with stage IIIb, IIIc or IV metastatic melanoma (AJCC 6th edition) with at least two lesions (lymph nodes relapse, or in transit metastasis, or unresectable cutaneous metastases, or visceral metastases except bone and brain metastases) including one easily accessible and no more than 2 lines of treatment of melanoma at the metastatic stage.
* Patients with a melanoma expressing a Braf V600 mutation can be included
* Measurable/assessable disease in 28 days which precede the first administration of the treatment
* A negative pregnancy test for women with childbearing potential
* Eastern Cooperative Oncology Group (ECOG) of 0-1, Karnofsky > 80%
* Laboratory results:

Haemoglobin ≥ 10 g/dl or ≥ 6,25 mmol/l; Neutrophils ≥ 1500/μl; Leukocytes ≥ 4000/μl; Lymphocytes ≥ 700/μl; Blood platelet ≥ 100.000/μl; Serum creatinine ≤ 1.5 x superior normal value or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula); Serum bilirubin ≤ 2.0 mg/dl or ≤ 34.2 mol/l; Total bilirubin ≤ 1.5 x superior normal value (except subjects with Gilbert Syndrome, who can have total bilirubin < 3mg/dL); Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2 x superior normal value; Lactate dehydrogenase (LDH) ≤ 1.5 x superior normal value

* Subjects affiliated to an appropriate health insurance
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception during the clinical trial. Furthermore WOCBP will be instructed to adhere to contraception for a period of 5 months after the last dose of Nivolumab.
* Men who are sexually active with WOCBP will be instructed to adhere to contraception during the clinical trial and for a period of 7 months after the last dose of Nivolumab.
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception.

Non inclusion Criteria:

* Brain or bone metastases
* Ocular melanoma
* Chemotherapy or radiotherapy within 4 weeks before baseline (6 weeks for nitroso-ureas and mitomycin C)
* Contraindication for the use of vasopressor agents
* For female: the patient is pregnant or breastfeeding or not using contraception
* For men: the patient is sexually active with WOCBP and not using contraception
* History or current manifestations of severe progressive heart disease (congestive heart failure, coronary artery disease, uncontrolled arterial hypertension, serious rhythm disorders or ECG signs of previous myocardial infarction)
* Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways except in the context of adjuvant or neoadjuvant
* History of allergies and Adverse Drug Reaction:

  * Hypersensitivity to human albumin, TIL excipient
  * Hypersensitivity to Nivolumab or related excipients
  * History of severe hypersensitivity reaction to any monoclonal antibody
  * Hypersensitivity to aldesleukin or to one of Proleukin excipients
* History of chronic autoimmune disease (Addison's disease, multiple sclerosis, Graves' disease, rheumatoid arthritis, systemic lupus erythematosus, etc…) except patient with active vitiligo or a history of vitiligo.
* History of uveitis or melanoma-associated retinopathy
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea.
* Presence of a second active cancer, with the exception of an in situ cervical cancer or a skin cancer different from the treated melanoma
* Unchecked thyroid dysfunction
* Any serious, acute or chronic illness id est active infection asking for antibiotics administration, coagulation's disorders, or any state asking for an unauthorized concomitant treatment described in this study
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of nonautoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Adults under a legal protection regime (guardianship, trusteeship, "sauvegarde de justice")

Exclusion Criteria:

* Positive viral serology for HIV (human immunodeficiency virus) 1/2, p24 Ag, HTLV1, HTLV2, B and C hepatitis or syphilis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment (adoptive T cell therapy associated to intravenous injections of Nivolumab) - Emergent Adverse Events | Within 12 months
  Clinical and biological criteria defined by the NCI (Common Terminology Criteria for Adverse Events - version 4.0, may 2009, http://ctep.cancer.gov)

SECONDARY OUTCOMES:
Efficacy of adoptive T cell therapy associated to intravenous injections of Nivolumab | At 12 months
  The overall tumor response will be evaluated according to the guidelines for Response Evaluation Criteria in Solid Tumors (RECIST1.1) and immune-related Response Criteria (irRC)
Duration of the clinical response | Within 12 months of follow-up
  Time interval between the evaluation of the first objective response and the first evaluation of disease progression or death, whichever occurs first
Progression-free survival | From the date of the first infusion of Nivolumab until the date of the first documented progression or the date of death from any cause, whichever came first, assessed up to 12 months
  Evaluation of the progression-free survival of patients treated with adoptive T cell therapy in combination with intravenous injections of Nivolumab
Overall survival | From the date of the first infusion of Nivolumab until the date of death, assessed up to 12 months
  Evaluation of the overall survival of patients treated with adoptive T cell therapy in combination with intravenous injections of Nivolumab
Specific immune monitoring n°1: Evaluate the fraction of TIL specific to Melan-A and MELOE-1 | Week 14 + week 18
  Evaluation of the fraction of TIL specific to two Human Leukocyte Antigen (HLA)-peptide complexes (Melan-A and MELOE-1)
Specific immune monitoring n°2: Evaluate the proportion of regulatory T cells | Day 0 (1st Nivolumab injection) + week 14 + week 18 + week 26 + week 38 + at the date of disease progression assessed up to 12 months
  Evaluation of the proportion of regulatory T cells
Specific immune monitoring n°3: Analyse the expression of tumor antigens | Week 10 + week 38
  Analysis of the expression of tumor antigens
Specific immune monitoring n°4: Analyse the expression of immunosuppressive cytokines | Week 10 + week 38
  Analysis of the expression of immunosuppressive cytokines
Specific immune monitoring n°5: Analyse the expression of indoleamine 2,3-dioxygenase (IDO) | Week 10 + week 38
  Analysis of the expression of IDO
Specific immune monitoring n°6: Analyse the expression of FoxP3 | Week 10 + week 38
  Analysis of the expression of FoxP3
Specific immune monitoring n°7: Analyse the expression of regulatory molecules | Week 10 + week 38
  Analysis of the expression of regulatory molecules
Specific immune monitoring n°8: Analyse the mutations of BRAF | Week 10 + week 38
  Analysis of BRAF mutations
Specific immune monitoring n°9: Analyse the mutations of Neuroblastoma Ras viral oncogene homolog (NRAS) | Week 10 + week 38
  Analysis of NRAS mutations
Specific immune monitoring n°10: Analyse the mutations of proto-oncogene ckit (cKit) | Week 10 + week 38
  Analysis of cKit mutations
Specific immune monitoring n°11: Determine the percentage of reactive T cells in the expanded cells | Week 10
  Produce tumor cell line and determine the percentage of reactive T cells in the expanded cells
Specific immune monitoring n°12: Determine the phenotype of the expanded T cells | Week 10
  Produce tumor cell line and determine the phenotype of the expanded T cells
Specific immune monitoring n°13: Test TIL reactivity | Week 10
  Produce tumor cell line and test TIL reactivity

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France